CLINICAL TRIAL: NCT01237275
Title: Development of A Technique to Predict Antidepressant Responsiveness in Depressive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D.,Ph.D., Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1999-10-14
Record Dates: First submitted 2010-11-01; First posted 2010-11-09 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Continuous Antidepressant Abuse; Adverse Reaction to Drug
Keywords: Pharmacogenomics; Prediction of Antidepressant Response; Depressed Patients
MeSH Terms: conditions — Depression; Drug-Related Side Effects and Adverse Reactions | interventions — Paroxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SSRI treated group (Experimental): SSRI treated group are depressive patients treated with fluoxetine, paroxetine or sertraline
  Interventions: Drug: SSRI treated group

INTERVENTIONS:
Drug: SSRI treated group — characterize in arm of a study (SSRI treated group)
  Other Names: fluoxetine_Prozac; paroxetine_Paxil, Seroxat; sertraline_Zoloft

SUMMARY:
First, the investigators examined the functional relevance of serotonin transporter polymorphisms by quantifying the activity of serotonin transporter in blood platelets of genotyped healthy volunteers and patients with major depression.

Second, the investigators studied response to SSRIs in relation to 5-HTTLPR genotype and also to the functional expression of 5-HTT in platelets.

DETAILED DESCRIPTION:
The purpose of this study is

1. to determine whether serotonin transporter genotypic or functional differences between depressive patients and normal controls were existed.
2. to determine the relationship between serotonin transporter polymorphisms and serotonin transporter functional expression.
3. to determine whether genomic or functional differences between drug responders and nonresponders predict the response of antidepressant

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were enrolled in the clinical trials program of hte Samsung Medical Center Geropsychiatry and Affective Disorder Clinics(Seoul, Korea). They received a semistructured diagnostic interview, the Samsung Psychiatric Evaluation Schedule. The affective disorder section of the Samsung Psychiatric Evaluation Schedule uses the Korean version of the structured clinical interview for the diagnostic and statistical manual of mental disorders, Fourth edition.
* interview with one more patient's family member for objective diagnosis and final diagnosis decision by agreements of two more psychiatric physicians

Exclusion Criteria:

* received psychotropic medication within 2 weeks of the study or fluoxetine within 4 weeks
* potential study participants for pregnancy, significant medical conditions, abnormal laboratory baseline values, unstable psychiatric features(eg.suicidal), history of alcohol of drug dependence, seizures, head trauma with loss of consciousness, neurological illness, or concomitant Axis I psychiatric disorder.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1999-10; Primary Completion 2003-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Antidepressant Response at 2,4,6 weeks | 6 weeks

SECONDARY OUTCOMES:
Biological value at 0 and 6 weeks | 6weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea